CLINICAL TRIAL: NCT01252940
Title: A Phase 3 Randomized, Open Label Study to Evaluate Switching From Regimens Consisting of a Ritonavir-boosted Protease Inhibitor and Two Nucleoside Reverse Transcriptase Inhibitors to Emtricitabine/Rilpivirine/Tenofovir Disoproxil Fumarate (FTC/RPV/TDF) Fixed-dose Regimen in Virologically Suppressed, HIV-1 Infected Patients
Brief Title: Study to Evaluate Switching From Regimens Consisting of a Ritonavir-boosted Protease Inhibitor (PI) and Two Nucleoside Reverse Transcriptase Inhibitors (NRTIs) to a Fixed-dose Tablet Containing Emtricitabine/Rilpivirine/Tenofovir DF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-264-0106; 2010-023178-37 (EudraCT Number)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-10

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; HIV; Treatment Experienced
MeSH Terms: interventions — Emtricitabine, Rilpivirine, Tenofovir Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FTC/RPV/TDF (Experimental): Participants will switch from their existing treatment regimen to the emtricitabine (FTC)/rilpivirine (RPV)/tenofovir disoproxil fumarate (TDF) single-tablet regimen (STR) at the beginning of the study.
  Interventions: Drug: FTC/RPV/TDF
- SBR/Delayed Switch (Experimental): Participants will stay on baseline regimen (SBR; their existing treatment regimen of PI+RTV plus 2 NRTIs) at the beginning of the study through Week 24, and may switch to the FTC/RPV/TDF STR (Delayed Switch) at the Week 24 visit.
  Interventions: Drug: FTC/RPV/TDF; Drug: PI; Drug: RTV; Drug: NRTIs

INTERVENTIONS:
Drug: FTC/RPV/TDF — Emtricitabine (FTC) 200 mg/rilpivirine (RPV) 25 mg/tenofovir disoproxil fumarate (tenofovir DF; TDF) 300 mg single-tablet regimen (STR) administered orally with a meal once daily (QD)
  Other Names: Complera®; Eviplera®
Drug: PI — Protease inhibitors (PIs) included amprenavir, atazanavir, darunavir, fosamprenavir, Kaletra (lopinavir/ritonavir, coformulated), ritonavir, and saquinavir. PIs were administered according to prescribing information.
  Arms: SBR/Delayed Switch
Drug: RTV — Ritonavir (RTV) was administered according to prescribing information.
  Arms: SBR/Delayed Switch
Drug: NRTIs — NRTIs included abacavir, emtricitabine, Combivir (lamivudine/zidovudine, coformulated), Epzicom (abacavir/lamivudine, coformulated), lamivudine, stavudine, tenofovir DF, Truvada® (emtricitabine/tenofovir DF, coformulated), and zidovudine. NRTIs were administered according to prescribing information.
  Arms: SBR/Delayed Switch

SUMMARY:
The purpose of this randomized, open-label, multicenter, active-controlled Phase 3b study is to evaluate the noninferiority of the emtricitabine/rilpivirine/tenofovir disoproxil fumarate (FTC/RPV/TDF) single-tablet regimen (STR; also referred to as fixed-dose regimen or fixed-dose tablet) relative to regimens consisting of a ritonavir-boosted protease inhibitor (PI+RTV) and two nucleoside reverse transcriptase inhibitors (NRTIs) in virologically suppressed, HIV-1 infected subjects. The FTC/RPV/TDF STR could offer an attractive treatment option to patients who wish to simplify dosing by reducing pill burden or to improve the tolerability of their treatment.

Participants will be randomized into 2 groups, the FTC/RPV/TDF STR group, in which participants will switch treatment regimens at the start of the study, and the Stay on Baseline Regimen (SBR)/Delayed Switch group, in which participants will remain on their baseline regimen during the first 24 weeks of the study (designed to provide an initial active control), and may switch to the FTC/RPV/TDF STR at the Week 24 visit.

After the 48-week study analysis period, participants may continue to receive the FTC/RPV/TDF STR per protocol before switching to a commercially available source.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form
* Receiving antiretroviral therapy with a ritonavir-boosted PI and two NRTIs continuously for ≥ 6 months preceding the screening visit
* Plasma HIV-1 RNA concentrations (at least two measurements) at undetectable levels for ≥ 6 months prior to the screening visit and HIV-1 RNA < 50 copies/mL at the screening visit
* On their first or second antiretroviral drug regimen; if on their second regimen, HIV-1 RNA ≤ 50 copies/mL required at the time of the first change in antiretroviral drugs, and no HIV RNA > 50 copies/mL measured at two consecutive time points after first achieving HIV RNA < 50 copies/mL
* No previous use of any approved or experimental nonnucleoside reverse transcriptase inhibitor (NNRTI) drug for any length of time
* Have a genotype prior to starting initial antiretroviral therapy and no known resistance to any of the study agents
* Normal ECG
* Hepatic transaminases (AST and ALT) ≤ 5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function (absolute neutrophil count ≥ 1,000/mm^3; platelets ≥ 50,000/mm^3; hemoglobin ≥ 8.5 g/dL)
* Serum amylase ≤ 5 x ULN (subjects with serum amylase > 5 x ULN eligible if serum lipase ≤ 5 x ULN)
* Adequate renal function (estimated glomerular filtration rate ≥ 70 mL/min according to the Cockcroft-Gault formula)
* Males and females of childbearing potential must agree to utilize highly effective contraception methods (two separate forms of contraception, one of which must have been an effective barrier method, or been nonheterosexually active, practice sexual abstinence, or have a vasectomized partner) from screening throughout the duration of the study period and for 30 days following the last dose of study drug.
* Age ≥ 18 years
* Life expectancy ≥ 1 year

Exclusion Criteria:

* A new AIDS-defining condition diagnosed within 30 days prior to screening except cluster of differentiation 4 (CD4) cell count and/or percentage criteria
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Proven or suspected acute hepatitis 30 days prior to study entry.
* Current alcohol or substance abuse judged by the Investigator to potentially interfere with subject compliance.
* History of malignancy within 5 years prior to study entry or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Active, serious infections requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Anticipated need to initiate contraindicated drugs during the study, including drugs not to be used with FTC, TDF, RPV; or subjects with known allergies to the excipients of FTC/RPV/TDF STR tablets or Truvada® tablets
* All investigational drugs
* Medications and use of herbal/natural supplements excluded or to be used with caution while participating in the study, including those not to be taken with Viread®, Emtriva®, Truvada, and Rilpivirine.
* Participation in any other clinical trial without prior approval from the sponsor was prohibited while participating in this trial
* Treatment with immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening, or expected to receive these agents or systemic steroids during the study
* History of liver disease, including Gilbert's Disease
* Any other clinical condition or prior therapy making the subject unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Flaherty, PharmD, Study Director — Gilead Sciences
Locations (111):
- United States (66):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Spectrum Medical Group, Phoenix, Arizona
  - Health for Life Clinic, PLLC, Little Rock, Arkansas
  - AIDS Healthcare Foundation-Research Center, Beverly Hills, California
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Center for Special Immunology, Costa Mesa, California
  - Kaiser Permanente, Hayward, California
  - The Living Hope Foundation, Long Beach, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Kaiser Permanente, Los Angeles, California
  - Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - Oasis Clinic, Los Angeles, California
  - Anthony Mills, MD Internal Medicine, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Alameda County Medical Center, Oakland, California
  - East Bay AIDS Center, Oakland, California
  - Stanford University, Palo Alto, California
  - University of California, Davis, Sacramento, California
  - Kaiser Permanente, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Metropolis Medical, San Francisco, California
  - Kaiser Permanente, San Francisco, California
  - Capital Medical Associates PC, Washington D.C., District of Columbia
  - Gary Richmond, MD, PA, Inc., Fort Lauderdale, Florida
  - Midway Immunology & Research Center, Ft. Pierce, Florida
  - The Kinder Medical Group, Miami, Florida
  - Care Resource, Miami, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - ValueHealthMD, LLC/IDOCF, Orlando, Florida
  - Wade, Barbara Private Practice, Pensacola, Florida
  - Barry M. Rodwick, M.D., Safety Harbor, Florida
  - University of South Florida - HIV Clinical Research Unit, Tampa, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Atlanta ID Group, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta (IDSA), Decatur, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - The Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Northstar Medical Center, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Lutherville, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Kansas City Free Health Clinic, Kansas City, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somer Point, New Jersey
  - Greiger Clinic, Mount Vernon, New York
  - Beth Israel Medical Center, New York, New York
  - The Aaron Diamond AIDS Research Center, New York, New York
  - ID Consultant, P.A., Charlotte, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - University of South Carolina, Columbia, South Carolina
  - Nicholaos Bellos, MD, PA, Dallas, Texas
  - Tarrant County Infectious Diseases Associates, Fort Worth, Texas
  - Garcia Family Medical Clinic, Harlingen, Texas
  - Therapeutic Concepts, P.A., Houston, Texas
  - Gordon E. Crofoot, MD, PA, Houston, Texas
  - Research Access Network, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research & Education-Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
- Austria (5):
  - Univ.-Kklinik fuer Innere Medizin III, Salzberg
  - LKH Graz West, Styria
  - 2.Interne Lungenabteilung Otto Wagner Spital, Vienna
  - Dept. of Dermatology, Div. of Immunology,, Vienna
  - Private Office, Vienna
- Belgium (3):
  - CHU Saint-Pierre University Hospital, Brussels
  - University Hospitals Leuven, Flemish Brabant
  - Universitaire Ziekenhuis Gent, Ghent
- Canada (5):
  - Downtown Infectious Disease Clinic - Univ of BC, Vancouver, British Columbia
  - Maple Leaf Research, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Clinique Medicale Du Quartier Latin, Montreal, Quebec
  - Winnipeg Regional Health Authority, Winnipeg
- France (9):
  - Hôpital Hôtel-Dieu, Lyon
  - Infectiologie - 7ème Ouest - CHU HOTEL DIEU, Nantes
  - Archet 1 CHU de Nice - 6ème Niveau - Infectiology, Nice
  - Department of Infectious Diseases, Saint-Louis hospital, Paris
  - Hôpital Saint Antoine, Servuce de Maladies Infectieuses, Paris
  - Bichat Hospital, Paris
  - Hopital Tenon, Paris
  - Maladies Infectieuses Dpt, Paris
  - Hôpital Haut Levêque, Pessac
- Germany (7):
  - EPIMED GmbH, Berlin
  - University of Bonn, Dep. of Internal Medicine I, HIV-Outpatient Clinic, Bonn
  - University of Cologne, Department of Internal Medicine, Cologne
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Infectio Research, Frankfurt
  - ICH Study Center Hamburg, Hamburg
  - University Medical Center Hamburg - Eppendorf, Hamburg
- Italy (5):
  - Ospedali Riuniti, Bergamo
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Azienda Ospedaliera San Paolo, Mallattie Infettive e Tropicali, Milan
  - Azienda Ospedaliera Luigi Sacco 1° Divisione Malattie Infettive, Milan
  - National Institute for Infectious Diseases "L. Spallanzani" IRCCS, Rome
- Clinical Research Puerto Rico, Inc., San Juan, Puerto Rico
- Spain (4):
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
- United Kingdom (6):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex
  - Barts and the London NHS Trust, London
  - Royal Free Hospital, London
  - Chelsea and Westminster Hospital Foundation Trust, London
  - Homerton Unversity Hospital, London
  - North Manchester General Hospital, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 110 sites in the North America and Europe. The first participant was screened on 17 November 2010. The last participant observation was on 28 October 2014.
Pre-assignment Details: 617 participants were screened.
Groups:
- FTC/RPV/TDF: Participants were randomized to switch from their existing treatment regimen to the emtricitabine (FTC)/rilpivirine (RPV)/tenofovir disoproxil fumarate (TDF) single-tablet regimen (STR) at the beginning of the study.
- SBR/Delayed Switch: Participants were randomized to stay on their existing treatment regimen (Stay on Baseline Regimen (SBR)) at the beginning of the study through Week 24, and switch to the FTC/RPV/TDF STR (Delayed Switch) at the Week 24 visit.
Period: Main Study Phase
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Started | 321 | 161
Completed 24 Weeks | 0 | 153 (152 participants switched regimens at Week 24.)
Completed | 295 | 149 (Discontinuations after switch: withdrawal by subject, 2; adverse event, 1; protocol violation, 1.)
Not Completed | 26 | 12
Not completed — Randomized but not treated | 4 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 6 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Subject Non-compliance | 1 | 1
Period: Extension Phase
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Started | 110 (FTC/RPV/TDF group: 110 participants completing the main study continued in extension phase.) | 49 (SBR/Delayed Switch Group: 49 participants completing the main study continued in extension phase.)
Completed | 100 | 46
Not Completed | 10 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 5 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Subject Non-compliance | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least one dose of study drug
Groups:
- FTC/RPV/TDF: Participants were randomized to switch from their existing treatment regimen to the FTC/RPV/TDF STR at the beginning of the study.
- Total: Total of all reporting groups
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch | Total
Number analyzed (Participants) | 317 | 159 | 476
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (9.2) | 43 (9.7) | 42 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 15 | 59
  Male | 273 | 144 | 417
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 31 | 82
  Not Hispanic or Latino | 264 | 128 | 392
  Unknown or Not Reported | 2 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White | 241 | 124 | 365
  Black or African American | 61 | 22 | 83
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 6 | 2 | 8
  Other | 6 | 9 | 15
Region of Enrollment [Number; unit: participants] — Four participants in the Switch to FTC/RPV/TDF group and 2 participants in the Stay on Baseline Regimen (SBR) group were randomized but were not treated. These subjects are included in the analysis of the baseline characteristic "Region of Enrollment" but are not included in the analysis of other baseline characteristics.
  participants
    Austria | 18 | 8 | 26
    Belgium | 15 | 13 | 28
    Canada | 15 | 10 | 25
    France | 29 | 14 | 43
    Germany | 31 | 12 | 43
    Italy | 16 | 10 | 26
    Puerto Rico | 16 | 2 | 18
    Spain | 15 | 5 | 20
    United Kingdom | 17 | 6 | 23
    United States | 149 | 81 | 230
Baseline HIV-1 RNA Category [Number; unit: participants]
  < 50 Copies/mL | 299 | 152 | 451
  50 to < 200 Copies/mL | 10 | 6 | 16
  200 to < 400 Copies/mL | 2 | 0 | 2
  400 to < 1000 Copies/mL | 2 | 0 | 2
  ≥ 1000 Copies/mL | 4 | 1 | 5
Stratification based on antiretroviral (ARV) use [Number; unit: participants]
  TDF or FTC/TDF + lopinavir (LPV)/ritonavir (RTV) | 82 | 49 | 131
  TDF or FTC/TDF + Other PI+RTV | 178 | 81 | 259
  Non-TDF-containing regimen + LPV/RTV | 15 | 9 | 24
  Non-TDF-containing regimen + Other PI+RTV | 42 | 20 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 (FDA Snapshot Analysis)
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the FDA snapshot analysis.
Time Frame: Week 24
Population: Full Analysis Set: participants who were randomized into the study and received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 317 | 159
percentage of participants | 93.7 | 89.9
Statistical Analysis 1: Comparison: FTC/RPV/TDF; Test type: Non-Inferiority or Equivalence — A 95% confidence interval (CI) for the difference between treatment groups in the percentages of virologic success was constructed using normal approximation. Noninferiority was assessed using a conventional 95% CI approach, with a noninferiority margin of 12%. It would be concluded that the FTC/RPV/TDF STR group was not inferior to the SBR group if the lower bound of the 2-sided 95% CI of the difference (FTC/RPV/TDF STR - SBR) in the response rate was greater than -12%; Mean Difference (Net) = 3.8, 95% CI 2-sided [-1.6 to 9.1]

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 (FDA Snapshot Analysis)
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the FDA snapshot analysis.
  By Week 48, participants FTC/RPV/TDF had received 48 weeks of treatment with FTC/RPV/TDF, while those in the SBR/Delayed Switch group had received only 24 weeks of treatment with FTC/RPV/TDF.
Time Frame: Week 48
Population: Participants in the Full Analysis Set in the FTC/RPV/TDF and the Delayed Switch to FTC/RPV/TDF groups were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 317 | 152
percentage of participants | 89.3 | 92.1

3. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4) Count Through Week 24
Description: The mean (SD) change in CD4 count was analyzed from baseline through Week 24.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set who had CD4 measurements at both baseline and Week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 298 | 148
cells/mm^3 | 20 (149.3) | 32 (158.1)

4. Secondary Outcome: Change From Baseline in CD4 Count Through Week 48
Description: The mean (SD) change in CD4 count was analyzed from baseline through Week 48.
  By Week 48, participants FTC/RPV/TDF had received 48 weeks of treatment with FTC/RPV/TDF, while those in the SBR/Delayed Switch group had received only 24 weeks of treatment with FTC/RPV/TDF.
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set who had CD4 measurements at both baseline and Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 287 | 143
cells/mm^3 | 10 (144.1) | -7 (154.1)

5. Secondary Outcome: Change From Baseline in Fasting Total Cholesterol Through Week 24
Description: The mean (SD) change from baseline in fasting total cholesterol (mg/dL) through Week 24 was analyzed.
Time Frame: Baseline to Week 24
Population: Participants in the Safety Analysis Set who had measurements for total cholesterol at both baseline and Week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 269 | 134
mg/dL | -25 (30.2) | -1 (25.9)

6. Secondary Outcome: Change From Baseline in Fasting Total Cholesterol Through Week 48
Description: The mean (SD) change from baseline in fasting total cholesterol (mg/dL) through Week 48 was analyzed.
  By Week 48, participants FTC/RPV/TDF had received 48 weeks of treatment with FTC/RPV/TDF, while those in the SBR/Delayed Switch group had received only 24 weeks of treatment with FTC/RPV/TDF.
Time Frame: Baseline to Week 48
Population: Participants in the Safety Analysis Set who had measurements for total cholesterol at both baseline and Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 265 | 139
mg/dL | -24 (32.9) | -24 (32.0)

7. Secondary Outcome: Change From Baseline in Fasting High-density Lipoprotein (HDL) Cholesterol Through Week 24
Description: The mean (SD) change from baseline in fasting HDL cholesterol (mg/dL) through Week 24 was analyzed.
Time Frame: Baseline to Week 24
Population: Participants in the Safety Analysis Set who had measurements for HDL cholesterol at both baseline and Week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 269 | 134
mg/dL | -4 (10.3) | -1 (8.2)

8. Secondary Outcome: Change From Baseline in Fasting HDL Cholesterol Through Week 48
Description: The mean (SD) change from baseline in fasting HDL cholesterol (mg/dL) through Week 48 was analyzed.
  By Week 48, participants FTC/RPV/TDF had received 48 weeks of treatment with FTC/RPV/TDF, while those in the SBR/Delayed Switch group had received only 24 weeks of treatment with FTC/RPV/TDF.
Time Frame: Baseline to Week 48
Population: Participants in the Safety Analysis Set who had measurements for HDL cholesterol at both baseline and Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 265 | 139
mg/dL | -2 (11.6) | -2 (8.0)

9. Secondary Outcome: Change From Baseline in Fasting Direct Low-density Lipoprotein (LDL) Cholesterol Through Week 24
Description: The mean (SD) change from baseline in fasting direct LDL cholesterol (mg/dL) through Week 24 was analyzed.
Time Frame: Baseline to Week 24
Population: Participants in the Safety Analysis Set who had measurements for direct LDL cholesterol at both baseline and Week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 270 | 134
mg/dL | -16 (25.6) | 0 (23.7)

10. Secondary Outcome: Change From Baseline in Fasting Direct LDL Cholesterol Through Week 48
Description: The mean (SD) change from baseline in fasting direct LDL cholesterol (mg/dL) through Week 48 was analyzed.
  By Week 48, participants FTC/RPV/TDF had received 48 weeks of treatment with FTC/RPV/TDF, while those in the SBR/Delayed Switch group had received only 24 weeks of treatment with FTC/RPV/TDF.
Time Frame: Baseline to Week 48
Population: Participants in the Safety Analysis Set who had measurements for direct LDL cholesterol at both baseline and Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 265 | 139
mg/dL | -16 (27.1) | -14 (26.8)

11. Secondary Outcome: Change From Baseline in Fasting Triglycerides Through Week 24
Description: The mean (SD) change from baseline in fasting triglycerides through Week 24 was analyzed.
Time Frame: Baseline to Week 24
Population: Participants in the Safety Analysis Set who had measurements for triglycerides at both baseline and Week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 269 | 134
mg/dL | -53 (110.0) | 3 (100.1)

12. Secondary Outcome: Change From Baseline in Fasting Triglycerides Through Week 48
Description: The mean (SD) change from baseline in fasting triglycerides through Week 48 was analyzed.
  By Week 48, participants FTC/RPV/TDF had received 48 weeks of treatment with FTC/RPV/TDF, while those in the SBR/Delayed Switch group had received only 24 weeks of treatment with FTC/RPV/TDF.
Time Frame: Baseline to Week 48
Population: Participants in the Safety Analysis Set who had measurements for triglycerides at both baseline and Week 48 were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch
Number analyzed (Participants) | 265 | 139
mg/dL | -64 (126.4) | -80 (141.1)

ADVERSE EVENTS:
Time Frame: Baseline through end of study (average 54 weeks)
Description: Safety Analysis Set: participants who were randomized and received at least one dose of study drug
Groups:
- FTC/RPV/TDF: The adverse events reported in this group are those that occurred at any time during the study in participants who were randomized to switch from their existing treatment regimen to the FTC/RPV/TDF STR at the beginning of the study.
- SBR/Delayed Switch (up to Week 24): The adverse events reported in this group are those that occurred in the first 24 weeks of the study in participants who were randomized to stay on their existing treatment regimen (Stay on Baseline Regimen (SBR)) at the beginning of the study and switch to the FTC/RPV/TDF STR (Delayed Switch) at the Week 24 visit.
- SBR/Delayed Switch (After Week 24): The adverse events reported in this group are those that occurred after Week 24 in participants who were randomized to stay on their existing treatment regimen (Stay on Baseline Regimen (SBR)) at the beginning of the study and switch to the FTC/RPV/TDF STR (Delayed Switch) at Week 24 visit.
Arm/Group | FTC/RPV/TDF | SBR/Delayed Switch (up to Week 24) | SBR/Delayed Switch (After Week 24)
Serious Adverse Events (participants affected / at risk) | 21/317 | 8/159 | 9/152
Other Adverse Events (participants affected / at risk) | 150/317 | 38/159 | 59/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TDF (N=317) | SBR/Delayed Switch (up to Week 24) (N=159) | SBR/Delayed Switch (After Week 24) (N=152)
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Shigella infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Substance-induced mood disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TDF (N=317) | SBR/Delayed Switch (up to Week 24) (N=159) | SBR/Delayed Switch (After Week 24) (N=152)
Diarrhoea (Gastrointestinal disorders) | 34 | 8 | 6
Nausea (Gastrointestinal disorders) | 13 | 5 | 10
Fatigue (General disorders) | 22 | 5 | 4
Nasopharyngitis (Infections and infestations) | 35 | 8 | 12
Upper respiratory tract infection (Infections and infestations) | 15 | 5 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 6 | 8
Headache (Nervous system disorders) | 31 | 6 | 6
Depression (Psychiatric disorders) | 18 | 4 | 6
Insomnia (Psychiatric disorders) | 21 | 3 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years